CLINICAL TRIAL: NCT05179629
Title: Effectiveness of M-Tapa Block for Postoperative Analgesia Management in Patients Underwent Laparoscopic Cholesistectomy
Brief Title: M-Tapa Block for Laparoscopic Cholesistectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 23
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Cholecystitis; Cholecystitis, Acute; Cholecystitis, Chronic
Keywords: Laparoscopic Cholesistectomy; M-Tapa Block; Postoperative Analgesia
MeSH Terms: conditions — Cholecystitis; Cholecystitis, Acute; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for laparoscopic cholesistectomy surgery will be included in the study. Patients will be randomly divided into two groups (Group M = M-TAPA group, Group C = Control group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant were blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M = M-TAPA group (Active Comparator): Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure. 100 mg tramadol will be performed for rescue analgesia.
  Interventions: Drug: M TAPA block
- Group C = Control group (No Intervention): Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. Postoperative patient evaluation will be performed by a pain nurse blinded to the procedure.
  Wound local anesthetic infiltration will be applied to the patients in the control group. 100 mg tramadol will be performed for rescue analgesia.

INTERVENTIONS:
Drug: M TAPA block — Under aseptic conditions, a high frequency linear probe will be placed on the costochondral angle in the sagittal plane. Then the probe will be slightly angled deeply to visualize the lower view of the perichondrium. We will perform M-TAPA with totally 30 ml (15 ml for each side) of %0,25 bupivacaine.
  Arms: Group M = M-TAPA group

SUMMARY:
Modified Perichondral Approach Thoracoabdominal Nerve (M-TAPA) block is a novel block that provides effective analgesia of the anterior and lateral thoracoabdominal walls during laparoscopic surgery, in which local anesthetic is applied only to the lower side of the perichondral surface. M-TAPA block is a good alternative for analgesia of the upper dermatome levels and the abdominal lateral wall, and may be an opioid-sparing strategy with satisfactory quality improvement in patients undergoing laparoscopic surgery.

DETAILED DESCRIPTION:
Modified Perichondral Approach Thoracoabdominal Nerve (M-TAPA) block is a novel block that provides effective analgesia of the anterior and lateral thoracoabdominal walls during laparoscopic surgery, in which local anesthetic is applied only to the lower side of the perichondral surface. M-TAPA block is a good alternative for analgesia of the upper dermatome levels and the abdominal lateral wall, and may be an opioid-sparing strategy with satisfactory quality improvement in patients undergoing laparoscopic surgery.

M-TAPA block provides analgesia at the level of T5-T11 in the abdominal region. Sonoanatomy is easy to visualize and the spread of local anesthetic can be easily seen. Analgesia occurs in several dermatomes thanks to the cephalocaudal spread of the local anesthetic solution. There are studies in the literature investigating the effectiveness of M-TAPA block for post-operative pain management in bariatric surgery.

In this study, the investigators aimed to evaluate the effectiveness of M-TAPA block for postoperative analgesia management after laparoscopic cholecystectomy surgery.Primary aim is to compare the postoperative pain scores (VAS), and secondary aim is to compare the postoperative rescue analgesic use and postoperative opioid consumption, and the side effects (allergic reaction, nausea, vomiting) associated with opioid use.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for laparoscopic cholesistectomy surgery under general anesthesia

Exclusion Criteria:

* Bleeding diathesis
* Receiving anticoagulant treatment
* Known local anesthetics and opioid allergy
* Infection of the skin at the site of the needle puncture
* Pregnancy or lactation
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores (Numerical Ratin Scala; 0=no pain, 10=the worst pain felt) | Postoperative 24 hours period
  Change from Baseline Pain Scores at Postoperative 24 hours.

SECONDARY OUTCOMES:
The need for rescue analgesia | Postoperative 24 hours period
  The amount of Tramodol using (mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Tulgar S, Senturk O, Selvi O, Balaban O, Ahiskalioglu A, Thomas DT, Ozer Z. Perichondral approach for blockage of thoracoabdominal nerves: Anatomical basis and clinical experience in three cases. J Clin Anesth. 2019 May;54:8-10. doi: 10.1016/j.jclinane.2018.10.015. Epub 2018 Oct 31. No abstract available. PMID 30388604
- [Background] Altiparmak B, Toker MK, Uysal AI, Turan M, Demirbilek SG. Reply to Tulgar et al.: Perichondral approach for blockage of thoracoabdominal nerves: Anatomical basis and clinical experience in three cases. J Clin Anesth. 2019 May;54:150-151. doi: 10.1016/j.jclinane.2018.12.005. Epub 2018 Dec 12. No abstract available. PMID 30553219
- [Background] Tulgar S, Selvi O, Thomas DT, Deveci U, Ozer Z. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides effective analgesia in abdominal surgery and is a choice for opioid sparing anesthesia. J Clin Anesth. 2019 Aug;55:109. doi: 10.1016/j.jclinane.2019.01.003. Epub 2019 Jan 9. No abstract available. PMID 30639940